CLINICAL TRIAL: NCT03448029
Title: RECCORD - Recording Courses of Vascular Diseases
Brief Title: RECCORD (Recording Courses of Vascular Diseases) Registry
Acronym: RECCORD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsche Gesellschaft für Angiologie, Gesellschaft für Gefäßmedizin e.V. (Other)
Responsible Party: Sponsor
Other Study IDs: RECCORD; DRKS00013585 (Registry Identifier: Deutsches Register Klinischer Studien); U1111-1209-6562 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2018-02-08; First posted 2018-02-27 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Vascular Diseases; Peripheral Artery Disease; Claudication; Critical Limb Ischemia; Diabetic Foot
Keywords: Vascular Diseases; Peripheral Artery Disease; Revascularisation; Outcome; Quality Management; Registry; Endovascular Intervention; Limb Amputation
MeSH Terms: conditions — Vascular Diseases; Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia; Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endovascular Patients: Patients undergoing endovascular interventions for symptomatic PAD

SUMMARY:
The RECording COurses of vasculaR Diseases registry (RECCORD registry) is an observational, prospective, multicentre, all-comers registry platform.

In the initial phase, patients referred for endovascular revascularization of peripheral artery disease (PAD) of the lower limbs will be prospectively included and followed up for at least one year.

At baseline, data on patients' demographic characteristics, comorbidities, previous peripheral interventions, medication, and clinical stage of PAD (Rutherford category), haemodynamic parameters, and procedural data including complications will be assessed.

Major adverse cardiac and limb events will be recorded at planned (at six and 12 months) and at any unplanned visits.

For details see NM Malyar et al., Rationale and design of the RECording COurses of vasculaR Diseases registry (RECCORD registry). Vasa. https://doi.org/10.1024/0301-1526/a000631

DETAILED DESCRIPTION:
For details see NM Malyar et al., Rationale and design of the RECording COurses of vasculaR Diseases registry (RECCORD registry). Vasa.

https://doi.org/10.1024/0301-1526/a000631

ELIGIBILITY:
Inclusion Criteria:

* any type of endovascular interventions for symptomatic PAD
* endovascular intervention for PAD of lower extremities, i.e. below the aorto-iliac bifurcation

Exclusion Criteria:

* patients undergoing hybrid-(surgical and endovascular) and/or surgical interventions for symptomatic PAD
* patients with a life expectancy of <6 months
* endovascular intervention for reasons other than symptomatic PAD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing endovascular revascularization for symptomatic peripheral artery disease of the lower extremities (located distal to the aorto-iliac bifurcation) will be included. The diagnosis of PAD will be derived from ICD-10 codes. Any endovascular procedure that is performed to a specifi c target lesion will be documented as operation and procedure codes (OPS codes) as they are defi ned by the German procedure classifi cation system (version 2015). Informed consent from each patient will be obtained prior to inclusion in the registry.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Outcome Quality after Revascularization: Complications | Up to 1 month
  Peri- and post-interventional complications (puncture-site complications & intervention-related complications over 30 days
Outcome Quality after Revascularization: Amputation | Up to 12 months
  Amputation-free survival (AFS)
Outcome Quality after Revascularization: Survival | Up to 12 months
  Survival at one year in CLI patients
Quality of Life: EQ-5D-5L questionnaire | At baseline, at 6 and 12 months
  EQ-5D-5L questionnaire to asses patient's health state and patient's self-rated health
Outcome Quality after Revascularization: Re-Intervention | Up to 12 months
  Number of re-interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum der Ludwig-Maximilians Universität, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Official RECCORD Homepage — https://www.reccord.de